CLINICAL TRIAL: NCT00674804
Title: Communicating a Cancer Diagnosis: Current Methods and Their Effects
Brief Title: Communicating a Cancer Diagnosis-Current Methods and Their Effects
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080127; 08-CC-0127; NCT00732667 (obsolete NCT alias)
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-07-16

CONDITIONS: Behavior; Cancer
Keywords: Communicating a Diagnosis; Cancer Diagnosis; Recurrence of Cancer; Initial Cancer Diagnosis
MeSH Terms: conditions — Behavior; Neoplasms

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will investigate how patients are informed of their cancer diagnosis or recurrence and will explore their experience in learning about the diagnosis. Specifically, it will:

* Distinguish methods of telling the diagnosis and identify its relationship to the type of cancer.
* Determine if the way a patient is informed of their diagnosis is associated with their level of satisfaction with the method of being informed.
* Identify who informs the patient of their diagnosis..
* Determine patient satisfaction with their diagnostic consult.
* Identify indicators of satisfaction with the diagnostic consultation.

Patients 18 years of age or older who are enrolled in or being screened for enrollment in a phase I, II or III clinical trial in the National Cancer Institute's Medical Oncology, Metabolism, Surgery or Neuro-Oncology branch may be eligible for this study.

Participants complete a 15-minute questionnaire that includes questions related to the how they were informed of their cancer diagnosis.

DETAILED DESCRIPTION:
Background:

- The goals of the study are to identify how a patient with a diagnosis of cancer is informed of their condition and to illuminate the way in which this information exchange occurs.

Objectives:

To distinguish, identify and determine:

* If the method by which a patient is informed of a diagnosis of cancer is associated with their level of satisfaction with that method of being informed
* Who tells the patient of their condition
* The methods used to inform a patient of their condition
* Prognostic indicators of high satisfaction within the diagnostic consult

Eligibility:

* Patients currently enrolled or being screened for enrollment for a phase I, II or III clinical trial at the National Cancer Institutes clinic center- specifically, within the following branch clinics: Medical Oncology, Metabolism, Surgery and Neuro-Oncology.
* Patient must be 18 years or older and be willing to participate in the study.

Design:

* Primary methodological practice is a self-administered questionnaire.
* Questionnaire to be completed by patient on same day that it is administered at NCI.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age greater than or equal to 18 years.
2. A patient diagnosed with cancer who is either currently enrolled in a protocol and receiving treatment or has come to NCI for consult and potential enrollment in a trial.
3. Ability to follow basic verbal instructions as observed by either an investigator of the study or as reported by a member of the patient's primary clinical team.
4. Patient must comprehend English, verbal and written, to be determined by the investigator distributing the questionnaire.

   -Patients with a hearing and/or visual impairment will be eligible to participate in the study if they so choose. Appropriate accommodations will be made.
5. Signed informed consent form.

EXCLUSION CRITERIA:

1. Patients that have cognitive impairments, such as mental challenges/retardation due to a congenital or developmental anomaly.

   a. Subjects with cognitive impairments are ineligible to participate in the study due to comprehension inabilities.
2. Patients who have developed dementia as a result of their disease or from an unspecified source are not eligible for participation due to both memory and overall cognitive deficits.
3. Patients that have multiple concurrent cancers are excluded from participation in this study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2008-04-24; Primary Completion 2009-07-16 (Actual); Study Completion 2009-07-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Maguire P, Pitceathly C. Key communication skills and how to acquire them. BMJ. 2002 Sep 28;325(7366):697-700. doi: 10.1136/bmj.325.7366.697. No abstract available. PMID 12351365
- [Background] Zachariae R, Pedersen CG, Jensen AB, Ehrnrooth E, Rossen PB, von der Maase H. Association of perceived physician communication style with patient satisfaction, distress, cancer-related self-efficacy, and perceived control over the disease. Br J Cancer. 2003 Mar 10;88(5):658-65. doi: 10.1038/sj.bjc.6600798. PMID 12618870
- [Background] Barnett MM. Does it hurt to know the worst?--psychological morbidity, information preferences and understanding of prognosis in patients with advanced cancer. Psychooncology. 2006 Jan;15(1):44-55. doi: 10.1002/pon.921. PMID 15750997